CLINICAL TRIAL: NCT04414670
Title: Clinical Outcome of Laparoscopic or Robotic Metroplasty for Uterine Isthmocele
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 109002-E
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-02

CONDITIONS: Laparoscopic or Robotic Metroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: C/S — laparoscopic or robotic metroplasty

SUMMARY:
To evaluate the clinical outcomes of conventional or robotic - laparoscopic metroplasty for uterine isthmocele with the aid of a bending probe.

ELIGIBILITY:
Inclusion Criteria:

* > 20 years of women
* uterine isthmocele status post laparoscopic or robotic metroplasty with a bent uterine sound

Exclusion Criteria:

* Those underwent traditional open surgery.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: uterine isthmocele status post laparoscopic or robotic metroplasty
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Change of prolonged menstrual bleeding condition | 10 years
  Symptoms improvement and perioperative complications

SECONDARY OUTCOMES:
Change of scar defect size | 10 years
  Symptoms improvement and perioperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No